CLINICAL TRIAL: NCT01552746
Title: From Acute to Chronic Postoperative Shoulder Pain in Patients for Elective Lobectomy
Acronym: FACTS2
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: Vejle Hospital (Other)
Responsible Party: Principal Investigator, Morten Rune Eckhardt, Afdelingslæge, Ph.d.-studerende, Odense University Hospital
Other Study IDs: FACTS2
Record Dates: First submitted 2012-03-02; First posted 2012-03-13 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Pain
Keywords: Postoperative shoulder pain; Persisting postoperative pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Shoulder pain is a well known problem after thoracical surgery. The pathogenesis of the pain is uncertain, but mainly a mix of referred pain and mechanical strain to the shoulder. It is believed to last a few days. Persisting shoulder pain after thoracical surgery is a problem 1 year after surgery, but it is unknown if it is related to acute postoperative shoulder pain.

The purpose of the study is to systematically describe postoperative shoulder pain after lobectomy and examine the time progress up to 1 year after surgery.

DETAILED DESCRIPTION:
Further study details are provided by Departement V, Odense University Hospital

ELIGIBILITY:
Inclusion Criteria:

* Patients for elective lobectomy
* 18 years or older at the day of the operation
* Satisfactory abilities to speak and read danish

Exclusion Criteria:

* Previous Thoracical Surgery.
* Patients with diseases in the nervous system.
* Patients with preoperative shoulder pain, neuropathies or sensory disturbances in the arm or shoulder.
* Patients who are reoperated in the thorax in the study period or any other body-region within the first 4 postoperative days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients, scheduled for elective lobectomy of the lung at Odense University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain | 12 months
Shoulder range of motion | 12 months
  Shoulder range of motion in: flexion, outward rotation, inward rotation, adduction

SECONDARY OUTCOMES:
Thoracical Pain | 12 months
Presence of allodynia and hyperalgesia on the shoulder on the operated side. | 1. postoperative day
  Presence of allodynia and hyperalgesia on the shoulder on the operated side, compared to the contralateral shoulder.
Quantitative sensory testing values on the shoulder | 12 months
  Quantitative sensory testing values in referred pain area compared to contralateral side and preoperative values.
  The following quantitative sensory tests are performed:
  Cold Detection Threshold,Warm Detection Threshold, Cold Pain Threshold, Heat Pain Threshold, Mechanical detection Threshold, Mechanical Pain Threshold, Mechanical Pain Sensitivity, Allodynia, Wind-Up Ratio, Vibration Detection Threshold, Pressure Pain Threshold
Hospital Anxiety and Depression Score | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Morten R Eckhardt, MD, Principal Investigator — Departement V of anesthesia and intensive care, Odense University Hospital
Locations (1):
- Departement V of anesthesia and intensive care, Odense University Hospital, Odense, Denmark